CLINICAL TRIAL: NCT02891772
Title: Carotid Artery Corrected Flow Time Measured by Ultrasonography as a Predictor of Hypotension After Induction of General Anesthesia
Status: Withdrawn | Type: Observational
Why Stopped: The investigator's workplace and department were changed so that the study could no longer be carried out.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2016-0606
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: General Anesthesia Induction for Elective Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hypotension after anesthetic induction group: Patients with hypotension after anesthetic induction
  Interventions: Procedure: ultrasonographic measurement of corrected flow time(FTc) in carotid artery

INTERVENTIONS:
Procedure: ultrasonographic measurement of corrected flow time(FTc) in carotid artery — Corrected carotid artery flow time is measured using 10-5 MHz linear probe on a portable ultrasound machine. On the two-dimensional image, the optimal image of the long-axis view is obtained at the left common carotid artery. The sample volume is placed on the center of the lumen, 2 cm proximal to the bulb, and a pulsed wave Doppler examination was performed. Then, cardiac cycle time and carotid flow time is measured. Carotid flow time is measured between the upstroke of the flow tracing and the dicrotic notch, and it is corrected for pulse rate by dividing flow time by the square root of the cardiac cycle time to calculate corrected carotid artery flow time (flow time/√cycle time). The blood pressure was taken before anesthetic induction and every two minutes after anesthetic induction till ten minutes after endotracheal intubation.

SUMMARY:
Hypotension often happens immediately after anesthetic induction. Particularly in 5-10 minutes after anesthetic induction it is reported to happen more frequently. Patients may have preexisting hypovolemia resulting from dehydration and impaired compensatory responses, which increase the risk. However, it is still challenging to assess intravascular volume status in spontaneously breathing patients before anesthetic induction. Recently, the measurement of corrected flow time in carotid artery was introduced as quite useful, simple and noninvasive for the evaluation of circulating blood volume. The aim of this study is to evaluate whether corrected carotid artery flow time as determined by ultrasonography in spontaneously breathing patients before general anesthesia can predict hypotension after induction.

ELIGIBILITY:
Inclusion Criteria:

• adult patients (19-80 years of age) who were scheduled to undergo elective surgery under general anesthesia

Exclusion Criteria:

* mean blood pressure < 70 mmHg before induction of general anesthesia
* Patients who have currently taken angiotensin-converting enzyme inhibitor
* Patients who have currently taken angiotensin receptor blocker
* the presence of carotid artery stenosis > 50%
* cardiac rhythm other than sinus
* unstable angina
* a left ventricular ejection fraction of < 40%
* severe vascular disease
* implanted pacemaker/cardioverter
* autonomic nervous system disorders
* anticipated difficult airway
* pregnancy

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were scheduled to undergo elective surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
corrected flow time (FTc) in carotid artery | 10 minutes before induction of general anesthesia.
  the area under the receiver operating characteristics curve of corrected flow time in carotid artery measured by ultrasonography to predict hypotension after anesthetic induction

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No